CLINICAL TRIAL: NCT06082739
Title: Effectiveness of Various Exercises in Managing Kyphosis
Brief Title: Managing Kyphosis With Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, David Skaggs, Director Spine Center, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002960
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Kyphosis
Keywords: Scheuermann's; thoracolumbar; postural; stretching; back
MeSH Terms: conditions — Kyphosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise group (Experimental): Patients perform stretching exercises daily.
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — Stretching exercises with and without a bolster, ball, or foam roller.

SUMMARY:
The primary objective of this study is to determine if stretching exercises as a conservative treatment option will correct kyphosis in postural and Scheuermann's kyphosis.

DETAILED DESCRIPTION:
Despite comprehensive documentation of surgical interventions in existing literature, the investigation into non-operative approaches for addressing hyperkyphosis or Scheuermann's kyphosis in the pediatric population has been investigated with inconsistent findings. Various outcomes have been observed with regard to the effectiveness of multiple brace treatment options, alongside recommendations for various physiotherapeutic approaches, either in conjunction with brace treatment or as standalone interventions.

However, there is no universally accepted consensus regarding the conservative management of kyphosis that simultaneously ensures substantial patient satisfaction and heightened bodily awareness. Notably, there have been no studies investigating the efficacy of stretching in the treatment of individuals with kyphosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 8 and older with postural or Scheuermann's kyphosis with >45° of kyphosis or >10° of thoracolumbar kyphosis from T11-L1 or other cases which seem to have excessive kyphosis.
* Parents of patients aged 17 and younger who are 18 and older and cognitively able to complete a survey will be included in the study as well.

Exclusion Criteria:

* Patients with congenital kyphosis or scoliosis greater than 30°.
* Parents of patients aged 17 and younger who are less than 18 years of age or cognitively unable to complete a survey will be excluded from the study.
* Any records flagged "break the glass" or "research opt out."

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Kyphosis angle | Enrollment, 6-month follow-up, 2-year follow-up
  Change in severity of kyphosis angle evaluated using radiographs

SECONDARY OUTCOMES:
Patient Satisfaction and Perception | Enrollment, 6-month follow-up, 2-year follow-up
  Patient Satisfaction and Perception measured via questionnaires
Parental Perception | Enrollment, 6-month follow-up, 2-year follow-up
  Parental Perception of kyphosis measured via questionnaires
Exercise Adherence | Enrollment, 6-month follow-up, 2-year follow-up
  Exercise Adherence measured via questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: David L Skaggs, MD, MMM, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Priftis KN, Hager J, Vlachou M, Anthracopoulos MB. Effects of bracing on lung function in idiopathic juvenile kyphosis. Pediatr Pulmonol. 2003 Feb;35(2):83-6. doi: 10.1002/ppul.10220. PMID 12526067
- [Background] Karavidas NS. Bracing for Adolescent Idiopathic Scoliosis (AIS) and Scheuermann Kyphosis: the issue of overtreatment in Greece. Scoliosis Spinal Disord. 2016 Oct 14;11(Suppl 2):30. doi: 10.1186/s13013-016-0095-6. eCollection 2016. PMID 27785469
- [Background] Mehdikhani M, Behtash H, Ganjavian MS, Khalaj N. Orthotic treatment of idiopathic hyperkyphosis with Milwaukee brace. J Back Musculoskelet Rehabil. 2016 Aug 10;29(3):515-9. doi: 10.3233/BMR-150651. PMID 26836834
- [Background] Pizzutillo PD. Nonsurgical treatment of kyphosis. Instr Course Lect. 2004;53:485-91. PMID 15116637
- [Background] Riddle EC, Bowen JR, Shah SA, Moran EF, Lawall H Jr. The duPont kyphosis brace for the treatment of adolescent Scheuermann kyphosis. J South Orthop Assoc. 2003 Fall;12(3):135-40. PMID 14577720
- [Background] Tsirikos AI, Jain AK. Scheuermann's kyphosis; current controversies. J Bone Joint Surg Br. 2011 Jul;93(7):857-64. doi: 10.1302/0301-620X.93B7.26129. PMID 21705553
- [Background] Elpeze G, Usgu G. The Effect of a Comprehensive Corrective Exercise Program on Kyphosis Angle and Balance in Kyphotic Adolescents. Healthcare (Basel). 2022 Dec 8;10(12):2478. doi: 10.3390/healthcare10122478. PMID 36554002